CLINICAL TRIAL: NCT03145922
Title: Epigenetic Regulation of Altered T-cell Immunity in Sarcoidosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Collaborators: University of California, San Francisco (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, Brian O'Connor, Assoc. Professor, National Jewish Health
Other Study IDs: 15-18171
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Sarcoidosis; Sarcoidosis, Pulmonary
MeSH Terms: conditions — Sarcoidosis; Sarcoidosis, Pulmonary | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Sarcoidosis
  Interventions: Other: Observational Study
- Healthy Controls
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — Observational study utilizing bronchoscopy, and imaging

SUMMARY:
Sarcoidosis is a multi-system granulomatous disorder that is triggered and influenced by gene-environment interactions. Although sarcoidosis predominantly affects the lungs in most cases, the clinical disease course is highly variable and any organ can be affected leading to end organ damage despite currently available therapeutics that unfortunately also have numerous and potentially devastating side effects. The environmental triggers of sarcoidosis are unknown but several occupational, environmental and infectious agents have been associated with sarcoidosis in susceptible hosts. Exposure to these triggers result in inflammation, characterized by activation of CD4+ T-cells, cytokine production, subsequent recruitment of other immune cells, and granuloma formation. Although several genetic markers have been associated with sarcoidosis, none fully explain individual susceptibility or clinical course variability, strongly implicating the environment and epigenetics. We have the ability to generate a map of the epigenetic histone modifications in immune cells via Chromatin Immuno-Precipitation coupled with next generation sequencing (ChIP-seq) and a map of transcriptome profiles via RNA-seq. The availability of histone and transcriptional signatures defining T cell activity in sarcoidosis will help identify the specific molecular programs affected by disease processes and can become the basis for future discovery of novel biomarker diagnostics in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 85
* Diagnosis of sarcoidosis confirmed by either biopsy or by manifestations consistent with acute sarcoidosis in absence of other known diagnosis.
* Have a suspected diagnosis of sarcoidosis and is scheduled to undergo a biopsy procedure to confirm a diagnosis of sarcoidosis.
* Able to tolerate and willing to undergo study procedures

Exclusion Criteria:

* Current cigarette smoking or smoking within six months prior to the study
* Currently or recently (<6months) on immunosuppressive therapy
* Pregnancy
* Patient inability to participate in the study, such as undergo venipuncture and or BAL

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with Sarcoidosis.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Epigenomic Signature of Sarcoidosis | 5 years
  Determine the epigenomic signature of specific histone post-translational modifications associated with CD4+ T cell skewing and activity in sarcoidosis at the site of organ involvement via Chromatin Immuno-Precipitation coupled with next generation sequencing (ChIP-seq) and bronchoalveolar lavage (BAL).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco (Parnassus), San Francisco, California, United States